CLINICAL TRIAL: NCT02065687
Title: A Randomized Phase II/III Study of Paclitaxel/Carboplatin/Metformin (NSC#91485) Versus Paclitaxel/Carboplatin/Placebo as Initial Therapy for Measurable Stage III or IVA, Stage IVB, or Recurrent Endometrial Cancer
Brief Title: Paclitaxel and Carboplatin With or Without Metformin Hydrochloride in Treating Patients With Stage III, IV, or Recurrent Endometrial Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOG-0286B; NCI-2013-02284 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s14-01068; GOG-0286B; GOG-0286B (Other: NRG Oncology); GOG-0286B (Other: CTEP); U10CA180830 (NIH); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IV Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: interventions — Carboplatin; Metformin; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (paclitaxel, carboplatin, metformin hydrochloride) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1, carboplatin IV over 30 minutes on day 1, and metformin hydrochloride PO BID (approximately every 10-12 hours apart) on days 1-21 (QD in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising metformin hydrochloride PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  In both arms, patients who achieve SD or PR and still have measurable disease at the completion of course 6 may continue to receive paclitaxel IV and carboplatin IV (with metformin hydrochloride or placebo) for an additional 4 courses at the discretion of the treating investigator.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Metformin Hydrochloride; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (paclitaxel, carboplatin, placebo) (Active Comparator): Patients receive paclitaxel IV and carboplatin IV as in Arm I. Patients also receive placebo PO BID (approximately every 10-12 hours apart) on days 1-21 (QD in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising placebo PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  In both arms, patients who achieve SD or PR and still have measurable disease at the completion of course 6 may continue to receive paclitaxel IV and carboplatin IV (with metformin hydrochloride or placebo) for an additional 4 courses at the discretion of the treating investigator.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Metformin Hydrochloride — Given PO
  Other Names: APO-Metformin; Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; Glucophage ER; Metformin HCl; Riomet; Siofor
  Arms: Arm I (paclitaxel, carboplatin, metformin hydrochloride)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo Administration — Given PO
  Arms: Arm II (paclitaxel, carboplatin, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II/III trial studies how well paclitaxel, carboplatin, and metformin hydrochloride works and compares it to paclitaxel, carboplatin, and placebo in treating patients with endometrial cancer that is stage III, IV, or has come back. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Metformin hydrochloride may help paclitaxel and carboplatin work better by making cancer cells more sensitive to the drugs. It is not yet known whether paclitaxel and carboplatin is more effective with or without metformin hydrochloride in treating endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of metformin (metformin hydrochloride) to the standard regimen of carboplatin and paclitaxel prolongs progression-free survival (PFS) in women with advanced or recurrent endometrial cancer. (Phase II) II. To determine if the addition of metformin to the standard regimen of carboplatin and paclitaxel prolongs overall survival (OS) in the same population if a phase III study is conducted. Both clinical trials (Phase II and III) will utilize OS as a primary endpoint if a phase III trial is opened.

SECONDARY OBJECTIVES:

I. To estimate the proportion of patients with objective response (response rate [RR]) in the population of patients with measurable disease by treatment.

II. To estimate the duration of response in the population of patients with measurable disease who respond by treatment.

III. To estimate overall survival (OS) and relative hazards of death for each treatment arm if the study stops after the phase II trial is completed. If the study continues with a phase III clinical trial, then PFS will be a secondary endpoint.

IV. To determine the nature, frequency and degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) for each treatment arm.

V. To estimate possible differences in RR, PFS, OS, and toxicity rates for the treatment regimens by the patients' level of obesity.

TERTIARY OBJECTIVES:

I. To test whether PIK3CA mutations/amplifications, PTEN mutations or PIK3R1/PIK3R2 mutations have a lower hazard of progression or death (PFS endpoint) among patients who are treated with metformin.

II. To test whether higher expression of MATE 2 is associated with a lower hazard of progression or death (PFS endpoint) among patients who are treated with metformin.

III. To explore the association of metabolic factors (i.e. body mass index [BMI], hip-to-waist ratio, diabetes status, hemoglobin A1c [HgbA1C], fasting insulin and glucose levels, homeostatic model assessment [HOMA] scores) with treatment response to metformin/paclitaxel/carboplatin, PFS, and OS.

IV. To test whether genomic profiles (i.e. PIK3CA mutations/amplifications, PTEN mutations or PIK3R1/PIK3R2 mutations) differ between the tumors of obese and non-obese endometrial cancer (EC) patients.

V. To correlate expression of key targets of the insulin/IGF-1/mTOR signaling pathway (p-IGF1R, p-S6 and p-4EBP-1) with treatment response to metformin/paclitaxel/carboplatin, PFS, OS and obesity status.

VI. To determine if the genetic variants of the metformin transporters correspond with treatment response to metformin/paclitaxel/carboplatin, PFS and OS.

VII. To estimate differences in physical functioning, physical activity, and fatigue between treatment arms.

VIII. To explore the association between metabolic factors (i.e., BMI, hip-to-waist ratio, diabetes status, HgbA1C, fasting insulin and glucose levels, HOMA scores) and physical functioning, physical activity, and fatigue.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours on day 1, carboplatin IV over 30 minutes on day 1, and metformin hydrochloride orally (PO) twice daily (BID) (approximately 10-12 hours apart) on days 1-21 (once daily [QD] in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising metformin hydrochloride PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel IV and carboplatin IV as in Arm I. Patients also receive placebo PO BID (approximately 10-12 hours apart) on days 1-21 (QD in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising placebo PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

In both arms, patients who achieve stable disease (SD) or partial response (PR) and still have measurable disease at the completion of course 6 may continue to receive paclitaxel IV and carboplatin IV (with metformin hydrochloride or placebo) for an additional 4 courses at the discretion of the treating investigator.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable stage III, measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial carcinoma

  * Histologic confirmation of the original primary tumor is required; patients with the following histologic epithelial cell types are eligible:

    * Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.)
* Measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than 1.4 mg/dl
* Bilirubin less than or equal to 1.5 x institutional/laboratory upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Patients must NOT have received prior chemotherapy or targeted therapy, including chemotherapy used for radiation sensitization for treatment of endometrial carcinoma
* Patients may have received prior radiation therapy for treatment of endometrial carcinoma; prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy; all radiation therapy must be completed at least 4 weeks prior to the first date of study therapy
* Patients may have received prior hormonal therapy for treatment of endometrial carcinoma; all hormonal therapy must be discontinued at least one week prior to the first date of study therapy
* Patients must be able to swallow and retain orally-administered medication
* Patients must have signed an approved informed consent and authorization permitting release of personal health information; individuals with impaired decision-making capacity are not eligible to participate on the study

Exclusion Criteria:

* Patients must NOT be taking metformin or have been on metformin in the past 6 months
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the last three years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or nursing; if patients are of reproductive age and have not undergone hysterectomy, they must use an effective contraceptive method for the duration of this study
* Any condition associated with increased risk of metformin-associated lactic acidosis; (e.g. congestive heart failure defined as New York Heart Association [NYHA] class III or IV functional status, history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2023-09-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L Bae-Jump, Principal Investigator — NRG Oncology
Locations (431):
- United States (431):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Tennessee Valley Gynecologic Oncology, Huntsville, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology Associates-Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Arizona Oncology Associates-Wilmot, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Westchester Medical Center, Valhalla, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, Wilkesboro, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-The Woodlands, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - Virginia Gynecologic Oncology, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride): Patients receive 175 mg/m2 paclitaxel IV over 3 hours on day 1, carboplatin AUC 5 IV over 30 minutes on day 1, and 850 mg metformin hydrochloride PO BID (approximately every 10-12 hours apart) on days 1-21 (QD in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising metformin hydrochloride PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Paclitaxel, Carboplatin, Placebo): Patients receive 175 mg/m2 paclitaxel IV and carboplatin AUC 5 IV as in Arm I. Patients also receive placebo PO BID (approximately every 10-12 hours apart) on days 1-21 (QD in course 1). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising placebo PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Started | 234 | 235
Completed | 234 | 235
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo) | Total
Number analyzed (Participants) | 234 | 235 | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 64 (9) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 235 | 469
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 214 | 223 | 437
  Unknown or Not Reported | 8 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 39 | 22 | 61
  White | 171 | 201 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Time until disease progression, death, or date of last contact. This study was originally designed as a phase II/III study. It passed the phase 2 threshold and started the phase 3; however, a phase 3 interim analysis stopped the trial for futility. Therefore, data available for Phase III may be identical to data reported for Phase II or Phase II/III combined.
Time Frame: From date of study entry to time of progression or death, whichever occurs first, assessed up to 5 years
Population: All patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
Months | 9.0 [8.4 to 10.5] | 8.5 [8.0 to 10.3]

2. Primary Outcome: Overall Survival (OS) (Phase II and III)
Description: The observed length of life from randomization into the study to death or the date of last contact. This study was originally designed as a phase II/III study. It passed the phase 2 threshold and started the phase 3; however, a phase 3 interim analysis stopped the trial for futility. Therefore, data available for Phase III may be identical to data reported for Phase II or Phase II/III combined.
Time Frame: From date of study entry to time of death or the date of last contact, assessed up to 5 years
Population: All patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
Months | 34.6 [28.0 to 50.1] | 30.4 [24.6 to 37.8]

3. Secondary Outcome: Proportion of Patients Responding to Therapy
Description: The proportion of patients who had a response (complete or partial) by RECIST 1.1. Measurable disease is defined by RECIST (version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI.
Time Frame: During study treatment, up to 5 years.
Population: Evaluable for response
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 164 | 171
percentage of patients | 61.6 [53.7 to 69.1] | 60.2 [52.5 to 67.6]

4. Secondary Outcome: Duration of Response by Treatment
Description: Duration of response until disease progression, death, or date last seen among patients who responded.
Time Frame: From the date of response to disease progression, death, or date last seen assessed up to 5 years
Population: Patients who responded
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 101 | 103
Months | 8.0 [6.3 to 9.4] | 8.0 [6.2 to 10.3]

5. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: The observed length of life from randomization into the study to death or the date of last contact. For response, only those patients who had measurable disease were included in an analysis of response. Non-measurable patients are included in the ITT analysis. This study was originally designed as a phase II/III study. It passed the phase 2 threshold and started the phase 3; however, a phase 3 interim analysis stopped the trial for futility. Therefore, data available for Phase III may be identical to data reported for Phase II or Phase II/III combined.
Time Frame: From date of study entry to time of death or the date of last contact, assessed up to 5 years.
Population: All patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
Months | 34.6 [28.0 to 50.1] | 30.4 [24.6 to 37.8]

6. Secondary Outcome: Progression Free Survival (PFS) (Phase III)
Description: Time until disease progression, death, or date of last contact. For response, only those patients who had measurable disease were included in an analysis of response. Non-measurable patients are included in the ITT analysis. This study was originally designed as a phase II/III study. It passed the phase 2 threshold and started the phase 3; however, a phase 3 interim analysis stopped the trial for futility. Therefore, data available for Phase III may be identical to data reported for Phase II or Phase II/III combined.
Time Frame: From date of study entry to time of progression or death, whichever occurs first, assessed up to 5 years
Population: All patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
Months | 9.0 [8.4 to 10.5] | 8.5 [8.0 to 10.3]

7. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 4
Description: Toxicities will be assessed by organ or organ system. For each category of toxicity, each patient will be evaluated by the worst grade experienced during the course of therapy. Data will be summarized by frequency and severity according to the regimen administered. The number of patients with a grade three or greater adverse event will be reported (by system organ class).
Time Frame: Up to 5 years
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
Participants
  Blood and lymphatic system disorders | 23 | 17
  Cardiac disorders | 2 | 2
  Ear and labyrinth disorders | 1 | 0
  Endocrine disorders | 0 | 0
  Eye disorders | 0 | 0
  Gastrointestinal disorders | 17 | 10
  General disorders administration site conditions | 5 | 6
  Immune system disorders | 0 | 1
  Infections and infestations | 14 | 10
  Injury, poisoning and procedural complications | 2 | 6
  Investigations | 38 | 28
  Metabolism and Nutrition Disorders | 8 | 18
  Musculoskeletal and connective tissue disorders | 1 | 3
  Neoplasms benign, malignant and unspecified | 1 | 0
  Nervous system disorders | 8 | 9
  Psychiatric disorders | 0 | 2
  Renal and urinary disorders | 1 | 5
  Reproductive system and breast disorders | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 7 | 4
  Skin and subcutaneous tissue disorders | 2 | 1
  Vascular disorders | 10 | 18

8. Secondary Outcome: Level of Obesity
Description: Obesity will be quantitative assessed by body mass index (BMI) and will be assessed for its predictive and prognostic significance. The interaction between BMI and metformin treatment will be examined with an interaction term in a Cox proportional hazards model.
Time Frame: Up to 5 years
Population: All patients
Measure: Number; unit: proportion of participants obese
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
Number analyzed (Participants) | 234 | 235
proportion of participants obese | 0.4957 | 0.4979
Statistical Analysis 1: Comparison: Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) vs Arm II (Paclitaxel, Carboplatin, Placebo); The interaction between BMI and metformin treatment will be examined with an interaction term in a Cox proportional hazards model. Historical data indicate that approximately 50% of people are obese (BMI>=30). For the purposes of examining the relationship, we will classify patients into two levels (high versus low) at the median BMI, which will increase the likelihood of detecting an interaction between metformin treatment and obesity; Test type: Equivalence — The null hypothesis is that there is no relationship between BMI and metformin treatment (i.e. the parameter associated with the interaction term of BMI * treatment is equal to 0); p = 0.9482, Regression, Cox; Cox Proportional Hazard = -0.01787, Standard Error of Mean 0.27472

9. Other Pre Specified Outcome: Metabolic Factor Levels
Description: Hip-to-waist ratio, diabetes status, hemoglobin A1c, fasting insulin glucose levels, and homeostatic model assessment scores will be assessed for their predictive and prognostic significance. Variables will be analyzed as continuous covariates (or as appropriate with transformations such as the logarithm) with Cox models or logistic regression.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidence of PIK3 Mutations/Amplifications
Description: PIK3CA mutations/amplifications and PIK3R1/PIK3R2 mutations will be examined for prognostic and predictive significance.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Expression of MATE 2
Description: Expression will be examined by immunohistochemistry with intensity of staining and the percentage of cells staining positive. From these statistics, an H-score will be calculated. Expression will be further dichotomized as high expression and low expression at the median to maximize the power of the study.
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Levels of Key Targets of the Metformin/mTOR Signaling Pathway
Description: Levels before and after treatment will be assessed for their predictive and prognostic significance.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients are followed for the occurrence of adverse events for five years.
Arm/Group | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) | Arm II (Paclitaxel, Carboplatin, Placebo)
All-Cause Mortality (participants affected / at risk) | 95/234 | 95/235
Serious Adverse Events (participants affected / at risk) | 46/234 | 53/235
Other Adverse Events (participants affected / at risk) | 222/234 | 222/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) (N=234) | Arm II (Paclitaxel, Carboplatin, Placebo) (N=235)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Colonic Perforation (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 0 | 2
Infusion Related Reaction (General disorders) | 2 | 0
Anaphylaxis (Immune system disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 0 | 1
Uterine Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 5
Lung Infection (Infections and infestations) | 4 | 1
Device Related Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1
Catheter Related Infection (Infections and infestations) | 1 | 1
Bronchial Infection (Infections and infestations) | 1 | 0
Biliary Tract Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Weight Loss (Investigations) | 2 | 0
Creatinine Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Leukemia Secondary To Oncology Chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Ischemia Cerebrovascular (Nervous system disorders) | 1 | 0
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Bladder Perforation (Renal and urinary disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Metformin Hydrochloride) (N=234) | Arm II (Paclitaxel, Carboplatin, Placebo) (N=235)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 168 | 154
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 5
Atrial Fibrillation (Cardiac disorders) | 3 | 2
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 9 | 13
Myocardial Infarction (Cardiac disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Restrictive Cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 7 | 7
Chest Pain - Cardiac (Cardiac disorders) | 3 | 1
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 8 | 16
Hearing Impaired (Ear and labyrinth disorders) | 5 | 5
Vestibular Disorder (Ear and labyrinth disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 3 | 3
Hypothyroidism (Endocrine disorders) | 0 | 4
Hyperthyroidism (Endocrine disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Watering Eyes (Eye disorders) | 1 | 2
Flashing Lights (Eye disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 2
Photophobia (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 23 | 21
Dry Eye (Eye disorders) | 2 | 3
Floaters (Eye disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 18 | 18
Dry Mouth (Gastrointestinal disorders) | 6 | 4
Colonic Perforation (Gastrointestinal disorders) | 1 | 0
Colonic Fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 100 | 111
Diarrhea (Gastrointestinal disorders) | 133 | 79
Cheilitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 75 | 62
Bloating (Gastrointestinal disorders) | 9 | 11
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 5 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Anal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal Fistula (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 57 | 58
Rectal Hemorrhage (Gastrointestinal disorders) | 4 | 5
Oral Dysesthesia (Gastrointestinal disorders) | 0 | 2
Mucositis Oral (Gastrointestinal disorders) | 21 | 27
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Ileal Obstruction (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 4
Abdominal Distension (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 126 | 125
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 16 | 11
Rectal Pain (Gastrointestinal disorders) | 2 | 0
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Fecal Incontinence (Gastrointestinal disorders) | 1 | 3
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 7 | 2
Ascites (Gastrointestinal disorders) | 6 | 4
Toothache (Gastrointestinal disorders) | 3 | 3
Dental Caries (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 5 | 5
Gastritis (Gastrointestinal disorders) | 0 | 2
General Disorders And Administration Site Conditio (General disorders) | 0 | 1
Pain (General disorders) | 33 | 27
Malaise (General disorders) | 4 | 4
Localized Edema (General disorders) | 3 | 5
Injection Site Reaction (General disorders) | 2 | 0
Infusion Site Extravasation (General disorders) | 3 | 2
Flu Like Symptoms (General disorders) | 8 | 3
Edema Trunk (General disorders) | 1 | 4
Non-Cardiac Chest Pain (General disorders) | 9 | 12
Edema Limbs (General disorders) | 45 | 37
Edema Face (General disorders) | 1 | 2
Fatigue (General disorders) | 174 | 151
Fever (General disorders) | 14 | 15
Gait Disturbance (General disorders) | 6 | 3
Chills (General disorders) | 6 | 14
Infusion Related Reaction (General disorders) | 17 | 16
Anaphylaxis (Immune system disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 14 | 12
Autoimmune Disorder (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 2 | 1
Upper Respiratory Infection (Infections and infestations) | 9 | 9
Tooth Infection (Infections and infestations) | 3 | 2
Vulval Infection (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 2 | 0
Skin Infection (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 3 | 5
Sepsis (Infections and infestations) | 7 | 5
Rhinitis Infective (Infections and infestations) | 0 | 1
Rash Pustular (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1
Papulopustular Rash (Infections and infestations) | 2 | 2
Otitis Externa (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 3 | 4
Kidney Infection (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 0 | 1
Conjunctivitis Infective (Infections and infestations) | 1 | 1
Vaginal Infection (Infections and infestations) | 4 | 2
Urinary Tract Infection (Infections and infestations) | 28 | 21
Catheter Related Infection (Infections and infestations) | 1 | 1
Bronchial Infection (Infections and infestations) | 2 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Biliary Tract Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 4 | 1
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 11 | 7
Wound Complication (Injury, poisoning and procedural complications) | 2 | 3
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 10 | 16
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 2
Weight Loss (Investigations) | 27 | 22
Weight Gain (Investigations) | 3 | 9
Platelet Count Decreased (Investigations) | 90 | 85
Lymphocyte Count Increased (Investigations) | 1 | 1
Lymphocyte Count Decreased (Investigations) | 19 | 19
Inr Increased (Investigations) | 0 | 1
Hemoglobin Increased (Investigations) | 0 | 1
Ggt Increased (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 25 | 25
Cholesterol High (Investigations) | 2 | 1
Neutrophil Count Decreased (Investigations) | 117 | 119
Blood Bilirubin Increased (Investigations) | 5 | 4
White Blood Cell Decreased (Investigations) | 134 | 133
Aspartate Aminotransferase Increased (Investigations) | 19 | 25
Alkaline Phosphatase Increased (Investigations) | 27 | 24
Alanine Aminotransferase Increased (Investigations) | 27 | 24
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 6
Hyponatremia (Metabolism and nutrition disorders) | 29 | 32
Hypomagnesemia (Metabolism and nutrition disorders) | 49 | 32
Hypokalemia (Metabolism and nutrition disorders) | 34 | 35
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 28 | 39
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 7 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 56 | 46
Hypercalcemia (Metabolism and nutrition disorders) | 12 | 14
Glucose Intolerance (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 14 | 18
Anorexia (Metabolism and nutrition disorders) | 71 | 65
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 36 | 42
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 45 | 48
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 4 | 9
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range Of Motion Decreased Lumbar Spine (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 24 | 24
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 24 | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 30 | 36
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 55
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Leukemia Secondary To Oncology Chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tremor (Nervous system disorders) | 4 | 2
Transient Ischemic Attacks (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 145 | 157
Peripheral Motor Neuropathy (Nervous system disorders) | 14 | 16
Paresthesia (Nervous system disorders) | 20 | 9
Neuralgia (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 9 | 10
Lethargy (Nervous system disorders) | 3 | 1
Ischemia Cerebrovascular (Nervous system disorders) | 1 | 0
Movements Involuntary (Nervous system disorders) | 1 | 1
Intracranial Hemorrhage (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 44 | 33
Facial Muscle Weakness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 27 | 25
Dysesthesia (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 6 | 0
Dizziness (Nervous system disorders) | 33 | 37
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1
Concentration Impairment (Nervous system disorders) | 1 | 1
Cognitive Disturbance (Nervous system disorders) | 4 | 1
Ataxia (Nervous system disorders) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 3
Psychosis (Psychiatric disorders) | 1 | 0
Personality Change (Psychiatric disorders) | 1 | 3
Restlessness (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 36 | 42
Hallucinations (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 30 | 30
Delirium (Psychiatric disorders) | 0 | 2
Confusion (Psychiatric disorders) | 3 | 8
Anxiety (Psychiatric disorders) | 24 | 38
Agitation (Psychiatric disorders) | 3 | 6
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 7 | 5
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 12 | 19
Urinary Tract Pain (Renal and urinary disorders) | 14 | 15
Urinary Frequency (Renal and urinary disorders) | 19 | 14
Urinary Fistula (Renal and urinary disorders) | 1 | 0
Renal Calculi (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 5 | 3
Hematuria (Renal and urinary disorders) | 7 | 14
Cystitis Noninfective (Renal and urinary disorders) | 1 | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 2
Bladder Spasm (Renal and urinary disorders) | 1 | 1
Bladder Perforation (Renal and urinary disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Vaginal Perforation (Reproductive system and breast disorders) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 3 | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 11 | 19
Vaginal Dryness (Reproductive system and breast disorders) | 3 | 2
Uterine Hemorrhage (Reproductive system and breast disorders) | 1 | 0
Perineal Pain (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 8 | 12
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 11 | 11
Vaginal Inflammation (Reproductive system and breast disorders) | 2 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 63 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 38
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 1
Scalp Pain (Skin and subcutaneous tissue disorders) | 3 | 4
Rash Acneiform (Skin and subcutaneous tissue disorders) | 11 | 18
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 11
Pain Of Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 27 | 24
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 3 | 4
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 12 | 11
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 146 | 131
Thromboembolic Event (Vascular disorders) | 20 | 28
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 3 | 1
Lymphedema (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 5 | 8
Hypertension (Vascular disorders) | 40 | 47
Hot Flashes (Vascular disorders) | 24 | 28
Hematoma (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT02065687/Prot_SAP_000.pdf